CLINICAL TRIAL: NCT01923428
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of AZD1722 for the Treatment of Constipation-Predominant Irritable Bowel Syndrome (IBS-C)
Brief Title: The Efficacy of AZD1722 in Constipation Predominant Irritable Bowel Syndrome (IBS-C)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5612C00001
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Constipation Predominant Irritable Bowel Syndrome
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5 mg BID (Experimental): AZD1722
  Interventions: Drug: AZD1722
- 20 mg BID (Experimental): AZD1722
  Interventions: Drug: AZD1722
- 50 mg BID (Experimental): AZD1722
  Interventions: Drug: AZD1722
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1722
  Other Names: RDX5791, Tenapanor
  Arms: 20 mg BID; 5 mg BID; 50 mg BID
Drug: Placebo
  Arms: Placebo

SUMMARY:
This phase 2, randomized, double blind, placebo-controlled, multi-center study will evaluate the safety and efficacy of three dose levels of AZD1722 in subjects with constipation predominant IBS (IBS-C) as defined by the ROME III criteria and who have active disease as determined during a two-week screening period. Subjects who qualify and are randomized into the study will receive 5, 20, or 50 mg of AZD1722 BID or placebo BID for 12 consecutive weeks. At the end of this treatment period, subjects will be followed for an additional 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females and males must agree to use appropriate methods of contraception or be sterile (with appropriate documentation)
* Subject is ambulatory
* Subject meets definition of IBS-C using Rome III Criteria for the Diagnosis of IBS with a history of <5 SBMs per week
* Subject meets Screening eligibility criteria (see below)
* A colonoscopy based on AGA guidelines; every 10 years at ≥ 50 years old, or the occurrence of any warning signs (i.e., unexplained weight loss, non-hemorrhoid blood in stools)
* Ability to communicate well with the Investigator and to comply with the requirements of the entire study, including an understanding of how to use the touch-tone telephone electronic diary.
* Written informed consent and a willingness to participate in the study as it is described.
* Daily access to a touch tone telephone.

Exclusion Criteria:

* Functional diarrhea as defined by Rome III criteria
* IBS with diarrhea (IBS-D), mixed IBS (IBS-M), or unsubtyped IBS as defined by Rome III criteria
* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the GI tract within 6 months prior to screening, or active disease within 6 months prior to screening. Including but not limited to cancer, inflammatory bowel disease, diverticulitis, duodenal ulcer, erosive esophagitis, gastric ulcer, pancreatitis (within 12 months of screening), cholelithiasis, amyloidosis, ileus, non-controlled GERD, gastrointestinal obstruction or carcinoid syndrome.
* Use of medications that are known to affect stool consistency (Prohibited Medications), including fiber supplements, anti-diarrheals, cathartics, antacids, opiates, prokinetic drugs, laxatives, enemas, antibiotics within 4 weeks of enrollment, probiotics (including probiotic yogurt); or salt or electrolyte supplements containing sodium, potassium, chloride, or bicarbonate formulations during the seven days prior to treatment; unless specified as rescue medication, and used accordingly.
* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematologic, neurologic, psychiatric or any disease that may interfere with the subject successfully completing the trial.
* The subject has a history or current evidence of laxative abuse (in the clinical judgment of the physician).
* Hepatic dysfunction (ALT [SGPT] or AST [SGOT] >2.5 times the upper limit of normal) or renal impairment (serum creatinine > 2mg/dL).
* Any evidence of or treatment of malignancy (other than localized basal cell, squamous cell skin cancer or cancer in situ that has been resected) within the previous year.
* Any surgery on the stomach, small intestine or colon, excluding appendectomy.
* Pregnant or lactating women.
* A major psychiatric disorder (DSM-III-R or DSM-IV) including major depression or other psychoses that has required hospitalization in the last 3 years. History of attempted suicide or uncontrolled bipolar disorder. Alcohol or substance abuse in the last year.
* Participation in other clinical trials within 1 month prior to Day -14 (beginning of screening period).
* If, in the opinion of the Investigator the subject is unable or unwilling to fulfill the requirements of the protocol or has a condition, which would render the results uninterpretable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, Ph.D., Study Director — Ardelyx, Inc.
Locations (4):
- United States (4):
  - Boulder, Colorado
  - Greensboro, North Carolina
  - Winston-Salem, North Carolina
  - Chattanooga, Tennessee

REFERENCES:
- [Derived] Lacy BE, Shin AS, Cangemi DJ, Yang Y, Zhao S, Rosenbaum DP. Tenapanor is associated with earlier and sustained symptom relief in IBS-C: a post hoc analysis. Therap Adv Gastroenterol. 2026 Jan 24;19:17562848251414831. doi: 10.1177/17562848251414831. eCollection 2026. PMID 41601848

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
Period: Overall Study
Arm/Group | 5 mg BID | 20 mg BID | 50 mg BID | Placebo
Started | 88 | 89 | 89 | 90
Completed | 69 | 77 | 78 | 80
Not Completed | 19 | 12 | 11 | 10
Not completed — Adverse Event | 8 | 6 | 3 | 3
Not completed — Withdrawal by Subject | 5 | 3 | 0 | 4
Not completed — Lost to Follow-up | 2 | 1 | 5 | 0
Not completed — Protocol Violation | 3 | 0 | 2 | 1
Not completed — Non Compliance to treatment | 1 | 2 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg BID | 20 mg BID | 50 mg BID | Placebo | Total
Number analyzed (Participants) | 88 | 89 | 89 | 90 | 356
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 84 | 82 | 84 | 81 | 331
  >=65 years | 4 | 7 | 5 | 9 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 77 | 79 | 77 | 309
  Male | 12 | 12 | 10 | 13 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 30 | 24 | 29 | 105
  Not Hispanic or Latino | 66 | 59 | 65 | 61 | 251
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 18 | 19 | 17 | 22 | 76
  White | 69 | 67 | 69 | 65 | 270
  More than one race | 1 | 0 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (5.65) | 28.5 (5.27) | 28.3 (4.87) | 28.7 (5.63) | 28.7 (5.36)

OUTCOME MEASURES:

1. Primary Outcome: Percent Complete Spontaneous Bowel Movement Responders vs Placebo
Description: Weekly complete spontaneous bowel movement resaponders defined as an increase of one or more bowel movement per week from baseline for 6 of the 12 weeks
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg BID | 20 mg BID | 50 mg BID | Placebo
Number analyzed (Participants) | 87 | 87 | 84 | 89
Participants | 35 | 38 | 51 | 30
Statistical Analysis 1: Comparison: 50 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 27

ADVERSE EVENTS:
Arm/Group | 5 mg BID | 20 mg BID | 50 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 2/88 | 1/89 | 0/89 | 1/90
Other Adverse Events (participants affected / at risk) | 10/88 | 13/89 | 15/89 | 4/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg BID (N=88) | 20 mg BID (N=89) | 50 mg BID (N=89) | Placebo (N=90)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal neoplasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg BID (N=88) | 20 mg BID (N=89) | 50 mg BID (N=89) | Placebo (N=90)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 11 (11) | 10 (10) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 2 (2) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days